CLINICAL TRIAL: NCT01730794
Title: A Comparative, Multicenter, Randomized, Controlled Study of Neurally Adjusted Ventilatory Assist (NAVA) vs. Conventional Lung Protective Ventilation in Patients With Acute Respiratory Failure
Brief Title: Neurally Adjusted Ventilatory Assist (NAVA) Study in Adults With Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, Professor of Anesthesia, Director of Respiratory Care Services, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012P002419
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Acute Respiratory Failure
Keywords: Acute Respiratory Failure; Mechanical Ventilation; NAVA; Lung protective ventilation; invasive ventilation; noninvasive ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Lung Protective Ventilation (Other): In this group, patients will be ventilated in either volume A/C, pressure A/C, pressure support, pressure regulated volume control or volume support based on the discretion of the medical team with TV 4-8 ml/kg PBW range and PP or pressure (control or support) level <30 cmH2O.
  Interventions: Other: Conventional Lung Protective Ventilation
- NAVA Ventilation Group (Other): In the NAVA group, NAVA level will be set initially at zero, then the maximum Edi will be determined as the average level over the next 3 to 5 breaths without ventilatory support or PEEP. The actual NAVA level will then be titrated by the clinician to achieve the following: 1) an Edi equal to approximately 50% of the maximum Edi, 2) an average tidal volume of between 4 to 8 ml/kg predicted body weight (PBW), and 3) an average respiratory rate between about 15 and 40 per minute. In addition, the trigger sensitivity should be set as sensitive as possible without causing auto-triggering and the maximum pressure limit in NAVA should be set at 40 cm H2O.
  Interventions: Other: NAVA ventilation

INTERVENTIONS:
Other: NAVA ventilation — Neurally adjusted ventilatory assist
  Arms: NAVA Ventilation Group
Other: Conventional Lung Protective Ventilation — conventional protective mechanical ventilation
  Arms: Conventional Lung Protective Ventilation

SUMMARY:
The purpose of this study is to compare a specific mode of artificial ventilation (help from a breathing machine) with other modes. This specific mode is called Neurally Adjusted Ventilatory Assist (NAVA) and is different from other modes as it uses direct signals from the diaphragm (breathing muscle) to help patients breathe. The investigators believe that using these signals, NAVA can determine the exact timing for patients' spontaneous breathing effort and delivers the artificial breath at the same time (in synchrony) with their own breath. Other modes (breathing methods) may cause asynchrony between the patient and the ventilator while delivering artificial breaths because of the way they operate. Asyncrony between patient and ventilator is a risk factor for increasing the length of artificial ventilation and number of related complications. The investigators would like to find out if NAVA performs better in establishing synchrony between patient and ventilator and as a result decreasing time for artificial ventilation and increasing better outcomes.

DETAILED DESCRIPTION:
Study Goal To compare the ability of NAVA vs. conventional lung protective ventilation in a multicenter, unblinded, randomized, controlled fashion to provide invasive ventilatory support during acute respiratory failure in adults who are expected to require ventilatory support for greater than 72 hours.

Hypothesis It is hypothesized that the use of NAVA compared to conventional lung protective ventilation will result in a decrease in the number of days of mechanical ventilation. It is further hypothesized that NAVA compared to conventional lung protective ventilation will result in a decrease in the length of weaning, the length of ICU and hospital stay, and mortality.

Primary Outcome

• Number of invasive ventilator free days.

Secondary Outcome

* Mortality
* Length of Invasive Ventilation in survivors
* Length of ICU and hospital stay
* Incidence of barotrauma (defined as the presence of any extra-pulmonary air that was not present at study enrollment).
* Ventilator associated pneumonia (development of a pneumonia 48 hrs after entry into the study).
* Development of ARDS (after enrollment into the study; defined as a rapid onset, a P/F<200 mmHg, and bilateral pulmonary infiltrates that are not of cardiac origin).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Hypoxemic or hypercapnic acute respiratory failure
* Intubation and mechanical ventilation
* Anticipated mechanical ventilation equal or longer than 72 hrs
* Mechanically ventilated less or equal to 5 days
* Able to spontaneously trigger the ventilator

Exclusion Criteria:

* moderate-to-severe acute respiratory distress syndrome
* Post-operative patient's normally requiring a short course of mechanical ventilation (for example most cardiac surgical patients)
* Unable to spontaneously breathe
* Need to provide controlled ventilation
* Poor short term prognosis (defined as a high risk of death in the next 3 months)
* Neuromuscular or neurologic disease
* Age < 18 years
* Patients with major esophageal, gastric and oral surgery
* Acute brain injury or elevated intracranial pressure (> 18 mmHg)
* Severe cardiac disease: New York Heart Association class 3 or 4 or acute coronary syndrome or persistent ventricular tachyarrhythmias.
* Pregnancy, must be confirmed by laboratory analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Number of invasive ventilator free days. | 28 days
  Number of days without mechanical ventilation, within the first 28 days of the study.

SECONDARY OUTCOMES:
Total length of mechanical ventilation in survivors (invasive plus noninvasive) | 90 days
  Total number of days of mechanical ventilation in ICU survivors.
ICU and hospital Mortality | 90 days
  Mortality during patient stay in the ICU and after being discharged from ICU
Incidence of barotrauma | 60 Days
  Number of diagnosed pneumothorax
Ventilator associated pneumonia | 60 Days
  Number of diagnosed Ventilator Associated Pneumonia
Development of Acute respiratory distress syndrome (ARDS) | 60 Days
  Number of patients developing ARDS
Length of ICU stay | 90 Days
  Total number of days of ICU stay.
Length of hospital stay | 90 Days
  Total number of days of Hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kacmarek, PhD, Principal Investigator — Massachusetts General Hospital; Jesus Villar, MD, PhD, Principal Investigator — Hospital Universitario Dr. Negrín, Las Palmas de Gran Canaria, Spain
Locations (14):
- Nanjing Zhongda Hospital Southeast University, Nanjing, China
- Spain (13):
  - Hospital Universitario NS de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital NS del Prado, Talavera de la Reina, Toledo
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clinico de Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Txagorritxu, Vitoria-Gasteiz, Álava

REFERENCES:
- [Derived] Villar J, Belda J, Blanco J, Suarez-Sipmann F, Anon JM, Perez-Mendez L, Ferrando C, Parrilla D, Montiel R, Corpas R, Gonzalez-Higueras E, Pestana D, Martinez D, Fernandez L, Soro M, Garcia-Bello MA, Fernandez RL, Kacmarek RM; NAVa In Acute respiraTORy failure (NAVIATOR) Network. Neurally adjusted ventilatory assist in patients with acute respiratory failure: study protocol for a randomized controlled trial. Trials. 2016 Oct 13;17(1):500. doi: 10.1186/s13063-016-1625-5. PMID 27737690